CLINICAL TRIAL: NCT05999513
Title: A Phase 1, Open-Label, Randomized, Single-Dose, 3-Treatment, 3-Way Crossover, Pharmacokinetic Study to Evaluate the Relative Bioavailability of AB521 Tablet and Capsule Formulations and the Effect of Food on the Pharmacokinetics of the Tablet Formulation in Healthy Adult Volunteers
Brief Title: A Relative Bioavailability Study and Food Effect Study of AB521 in Healthy Adult Volunteers
Acronym: ARC-28
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARC-28
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
Keywords: AB521; casdatifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Casdatifan - Sequence ABC (Experimental): Participants will sequentially receive casdatifan capsules fasted (Treatment A), followed by casdatifan tablets fasted (Treatment B), followed by casdatifan tablets fed (Treatment C)
  Interventions: Drug: casdatifan
- Casdatifan - Sequence BCA (Experimental): Participants will sequentially receive Treatment B, followed by Treatment C, then Treatment A
  Interventions: Drug: casdatifan
- Casdatifan - Sequence CAB (Experimental): Participants will sequentially receive Treatment C, followed by Treatment A, then Treatment B
  Interventions: Drug: casdatifan

INTERVENTIONS:
Drug: casdatifan — Administered as specified in the treatment arm
  Other Names: AB521

SUMMARY:
The primary purpose of this study is to compare the single-dose pharmacokinetics (PK) of casdatifan tablet versus the casdatifan capsule, and to evaluate the effect of food on the single-dose PK of casdatifan tablet in healthy adult volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on volunteer self-reporting
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilogram (kg)/square meter (m^2) at the screening visit, with body weight ≥ 45 kg
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and ECGs, as deemed by the study physician
* Able to swallow multiple capsules and tablets
* Has adequate peripheral venous access

Key Exclusion Criteria:

* Has active neoplastic disease or history of neoplastic disease within 5 years of the screening visit (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care)
* Has abnormal liver enzyme test results or hematology values at the time of enrollment
* Has a history of additional risk factors for Torsades de pointes (example: heart failure, hypokalemia, family history of Long QT Syndrome)
* Malabsorption condition that would alter the absorption of orally administered medications at the discretion of the study physician
* Participation in another clinical study within 90 days or within 5 half-lives (if known), prior to the first dosing, whichever is longer. The 90-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Drug Concentration-Time Curve (AUC) | Predose, Up to 168 hours postdose
Maximum Concentration (Cmax) | Predose, Up to 168 hours postdose
Time to Maximum Concentration (Tmax) | Predose, Up to 168 hours postdose
Terminal Half-Life Time (t1/2) | Predose, Up to 168 hours postdose
Apparent Total Plasma Clearance (CL/F) | Predose, Up to 168 hours postdose
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) | Predose, Up to 168 hours postdose

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: Description ARC-28 - Public website — https://trials.arcusbio.com/study/?id=ARC-28